CLINICAL TRIAL: NCT03109249
Title: Pharmacokinetic Study of SPARC1613 and reference1613 in Subjects With Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLR_16_13
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Recurrent or Metastatic Breast Cancer
MeSH Terms: conditions — Recurrence; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SPARC1613 (Experimental): Intravenous administration of SPARC1613
  Interventions: Drug: Reference1613
- Reference 1613 (Active Comparator): Intravenous administration of Reference1613
  Interventions: Drug: SPARC1613

INTERVENTIONS:
Drug: SPARC1613 — Single intravenous infusion of 260 mg/m2 of SPARC1613 delivered over 25 minutes in either of two periods (Period 1 or 2)
  Arms: Reference 1613
Drug: Reference1613 — Single intravenous infusion of 260 mg/m2 of Reference1613 delivered over 30 minutes in either of two periods (Period 1 or 2)
  Arms: SPARC1613

SUMMARY:
SPARC1613 is chemotherapeutic agent with a wide spectrum of anti-tumor activity. It is used extensively in the treatment of advanced carcinomas of the breast, ovaries, lung, and other solid tumors.This is pharmacokinetic study of SPARC1613 and Reference1613.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate level of test medication with respect to time in the body, and safety when compared with the reference medication Subject will be randomly assigned to receive an intravenous infusion of either SPARC1613 delivered over 25 (±1) minutes or Reference1613 delivered over 30 (±1) minutes

ELIGIBILITY:
Inclusion Criteria:

* The subject has given written, informed consent and is available for the duration of study
* Histologically or cytologically confirmed diagnosis of breast cancer
* Male or female aged ≥ 18 years
* Females subjects of child-bearing potential must have a negative urine pregnancy test
* Female subjects must be non-lactating and non-breastfeeding
* Subject must be willing and able to comply with scheduled visits, treatment plan and laboratory testing

Exclusion Criteria:

* Known hypersensitivity to either of the study drugs or their excipients
* Inability to undergo venipuncture and/or tolerate venous access
* Pre-existing clinically significant peripheral neuropathy
* Positive laboratory exclusion test (HIV, HBsAg, or HCV)
* Treatment with investigational agents or participation in clinical trial within 30 days of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-01-14 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Pre-dose,post dose upto 3 days

OTHER OUTCOMES:
Adverse events | First dose of trial drug to one month after last dose.
  Adverse events encountered following dosing with SPARC1613 and Reference1613 will be recorded as per CTCAE4.03

CONTACTS AND LOCATIONS:
Locations (24):
- India (24):
  - SPARC Site 40, Visakhapatnam, Andhra Pradesh
  - SPARC Site 20, Ahmedabad, Gujarat
  - SPARC site 39, Ahmedabad, Gujarat
  - SPARC site 38, Karamsad, Gujarat
  - SPARC Site 27, Surat, Gujarat
  - SPARC Site 35, Surat, Gujarat
  - SPARC Site 24, Vadodara, Gujarat
  - SPARC Site 13, Bangalore, Karnataka
  - SPARC site 41, Bangalore, Karnataka
  - SPARC Site 28, Bangalore, Karnataka
  - SPARC Site 22, Belagavi, Karnataka
  - SPARC Site 7, Mangalore, Karnataka
  - SPARC Site 25, Aurangabad, Maharashtra
  - SPARC Site 23, Aurangabad, Maharashtra
  - SPARC Site 2, Mumbai, Maharashtra
  - SPARC Site 12, Nagpur, Maharashtra
  - SPARC site 34, Nashik, Maharashtra
  - SPARC Site 37, Nashik, Maharashtra
  - SPARC Site 18, Pune, Maharashtra
  - SPARC Site 4, Pune, Maharashtra
  - SPARC Site 9, Aurangabad, Marashtra
  - SPARC Site 15, Khordha, Odisha
  - SPARC site 42, Chennai, Tamil Nadu
  - SPARC Site 32, Madurai, Tamil Nadu

IPD SHARING:
Plan to Share IPD: No